CLINICAL TRIAL: NCT07200271
Title: Surgical Management of Lateral Ankle Instability: Modified Broström-Gould Versus Arthroscopic Allograft Reconstruction of the Anterior Talofibular and Calcaneofibular Ligaments. A Randomized Stratified Clinical Trial.
Brief Title: Surgical Management of Lateral Ankle Instability: Modified Broström-Gould Versus Arthroscopic Allograft Reconstruction of the Anterior Talofibular and Calcaneofibular Ligaments.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Francisco de Vitoria (Other)
Collaborators: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Responsible Party: Principal Investigator, Juan Chans Veres, Attending Physician, Foot and Ankle Unit, Department of Orthopaedic Surgery, Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: INEST2025
Record Dates: First submitted 2025-09-16; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Ankle Sprain
Keywords: ALLOGRAFT; INSTABILITY; ANKLE; LIGAMENT
MeSH Terms: conditions — Ankle Injuries | interventions — Conversion to Open Surgery

STUDY DESIGN:
Intervention Model Description: This is a randomized clinical trial with two parallel treatment arms, stratified by age and functional demand. One arm will undergo one of the reference surgical interventions for the treatment of chronic lateral ankle instability: the modified open Broström-Gould procedure. The other arm will undergo a more recently developed surgical intervention supported by studies with favorable outcomes: arthroscopic reconstruction of the anterior talofibular ligament and the calcaneofibular ligament.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open surgery arm (Active Comparator): Open surgery consists of the modified Broström-Gould technique, which allows for the reconstruction of damaged ligaments using the patient's own tissues through an incision on the lateral side of the fibula.
  Interventions: Procedure: Open surgery
- Arthroscopic surgery (Active Comparator): Arthroscopic reconstruction with allograft is a surgery in which a tendon (generally from a tissue bank) is used to reconstruct the ligaments. This technique is performed through small incisions using arthroscopy
  Interventions: Procedure: Arthroscopic reconstruction surgery

INTERVENTIONS:
Procedure: Arthroscopic reconstruction surgery — Arthroscopic reconstruction with allograft, in which a tendon (generally from a tissue bank) is used to reconstruct the ligaments. This technique is performed through small incisions using arthroscopy.
  Arms: Arthroscopic surgery
Procedure: Open surgery — Open surgery consists of the modified Broström-Gould technique, which allows for the reconstruction of damaged ligaments using the patient's own tissues through an incision on the lateral side of the fibula. This technique has shown satisfactory functional results.
  Arms: Open surgery arm

SUMMARY:
Primary Objective:

To clarify whether arthroscopic reconstruction with allograft provides tangible benefits over the modified open Broström-Gould technique, or if both are equivalent in efficacy and safety. The clinical AOFAS scale will be used for assessment.

Secondary Objectives:

To determine if there are differences in health outcomes and patient-perceived pain using the specific SP-36 scale and verbal numeric rating scale (VNRS). Additionally, to assess differences in postoperative complication rates and time to return to daily life activities between the two surgical techniques.

Study Design:

Prospective, randomized, controlled clinical trial with two parallel groups stratified by age and functional demand.

Condition or Disorder Being Studied:

Chronic lateral ankle instability.

Study Population and Sample Size:

The target population includes subjects diagnosed with chronic lateral ankle instability. The study population consists of patients diagnosed in the Orthopedics consultations at Hospital Infanta Elena who meet the inclusion and exclusion criteria. Based on sample size calculations, a total of 36 patients will be recruited. However, due to the prospective nature and stratification by epidemiological and functional variables, the sample size may be increased to ensure comparable groups in each stratum.

Study Timeline and Estimated Completion Date:

The study is expected to begin in the third quarter of 2025. Recruitment is estimated to last 24 months, with a follow-up period of 12 months, for a total duration of 3 years, ending in the third quarter of 2028.

ELIGIBILITY:
Inclusion Criteria:

Mandatory criteria (all must be marked "yes" in a drop-down tab):

* Age >18 years
* Subjective sensation of instability
* Pathological anterior drawer and varus tilt compared to the contralateral side
* Magnetic resonance imaging showing lesion of the anterior talofibular ligament (ATFL)

Specific criteria (must meet at least one, but can meet several, multiple choice option):

* BMI >30
* High athletic demand (regularly participates in pivoting sports)
* Ligamentous hyperlaxity (Beighton score >8)
* First sprain more than 2 years ago
* More than 5 sprains per year
* Subfibular ossicle >1 cm
* MRI with ATFL showing high T2 signal
* MRI showing disruption/absence of ATFL

Exclusion Criteria:

* History of previous ankle surgery
* Tibiotalar osteoarthritis or presence of chondral lesions on magnetic resonance imaging
* Active infections
* Contraindications for surgery
* Pregnancy
* Lactation
* Known allergy to bovine collagen
* Autoimmune connective tissue disease
* Active oncological process

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Clarify whether arthroscopic reconstruction with allograft provides tangible benefits over the modified open Broström-Gould technique, or if both are equivalent in efficacy and safety. | From surgery to the end of the follow up at 12 months after surgery
  Clarify whether arthroscopic reconstruction with allograft provides tangible benefits over the modified open Broström-Gould technique, or if both are equivalent in efficacy and safety. For this purpose, the clinical AOFAS (American Orthopedics Foot and Ankle Score) score will be used. The minimum value for the AOFAS score is 0 and the maximum value is 100. Higher scores on the AOFAS scale indicate a better outcome, meaning less pain, better function, and improved alignment.

SECONDARY OUTCOMES:
Determine whether there are differences in health outcomes | From surgery to the end of the follow up at 12 months after surgery
  Determine whether there are differences in health outcomes using the specific SP-36 (Short Form Health Survey) scale, is a 36-item questionnaire designed to measure health-related quality of life, it measures eight items: physical functioning, role limitations due to physical health, bodily pain, general health perceptions, vitality (energy/fatigue), social functioning, role limitations due to emotional problems and mental health. The score goes from 0 (worst health status) to 100 (best health status).
Determine whether there are differences in patient-perceived pain | From surgery to the end of the follow up at 12 months after surgery
  Determine whether there are differences in patient-perceived pain by using verbal numerical rating scale (VNRS). This score is widely used tool for assessing pain intensity, it measures pain from 0 (no pain) to 10 (worst paing imaginable).
Determine whether there are differences between both groups in the rate of postoperative complications. | From surgery to the end of the follow up at 12 months after surgery
  Determine whether there are differences between both groups in the rate of postoperative complications, defined as: Delay or absence of surgical wound healing, superficial infection, deep infection, recurrence or persistence of instability, sural nerve and superficial peroneal nerve neuropathy and complex regional pain syndrome. They are all qualitative variables. They will be expressed in the categories: yes or no.
Determine whether there are differences in time to return to normal life between the two surgical techniques. | From surgery to the end of the follow up at 12 months after surgery
  Determine whether there are differences in the time to return to normal life between the two surgical techniques. To do this, we will compare both groups in terms of time expressed in days.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Chans Veres, MD-PhD, Principal Investigator — Hospital Universitario Infanta Elena
Locations (1):
- Hospital Universitario Infanta Elena, Valdemoro, Madrid, Spain